CLINICAL TRIAL: NCT03628131
Title: Safety and Efficacy of Combination Chemotherapy With Pazopanib in Children and Adolescents With Relapsed/Refractory Solid Tumors
Brief Title: Combination Chemotherapy With Pazopanib in Children and Adolescents With Relapsed/Refractory Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-11-147
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Relapsed Pediatric Solid Tumor; Refractory Pediatric Solid Tumor
MeSH Terms: interventions — pazopanib; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pazopanib + conventional chemotherapy (Experimental): Conventional chemotherapy (Ifosfamide, carboplatin, etoposide) with Pazopanib
  Interventions: Drug: Pazopanib; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Pazopanib — Conventional chemotherapy (Ifosfamide, carboplatin, etoposide) with Pazopanib
Drug: Ifosfamide — Conventional chemotherapy (Ifosfamide, carboplatin, etoposide) with Pazopanib
Drug: Carboplatin — Conventional chemotherapy (Ifosfamide, carboplatin, etoposide) with Pazopanib
Drug: Etoposide — Conventional chemotherapy (Ifosfamide, carboplatin, etoposide) with Pazopanib

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of combination chemotherapy with Pazopanib in pediatric patients with relapsed/refractory solid tumor

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory/relapsed solid tumor (Stable or progressive disease after 1st-line treatment or relapse)
* Patients previously enrolled to "Genomic diagnosis of pediatric tumors by NGS (IRB No. SMC 2015-11-053)"

Exclusion Criteria:

* Patients who had high-dose chemotherapy and autologous stem cell transplantation previously
* Patients with organ dysfunction as follows (creatinine elevation ≥ 1.5 x upper limit of normal (ULN), ejection fraction <40%, significant arrhythmia or conduction disturbance)
* Patients who are not eligible to have scheduled treatment due to the other significant impaired organ function
* Patients with active bleeding
* Patients who are taking strong CYP3A4 inhibitors, QTc-prolonging drugs, antithrombotic agents, or anti-platelet agents
* Pregnant or nursing women
* Patients who can not swallow the pill

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Pazopanib in combination chemotherapy | 42 days
  Definition of dose-limiting toxicity (DLT)
  * Hematologic DLT: delayed recovery of ANC/platelets > 42 days
  * Grade 3 creatinine elevation, proteinuria, hyperbilirubinemia, bleeding
  * Grade 2 arterial thrombosis
  * Any grade 4 toxicities except hematologic toxicities

SECONDARY OUTCOMES:
Rate of tumor response (neuroblastoma) | 4 weeks
  * as assessed by International Neuroblastoma Response
  * Primary tumor: CT and/or MRI; MIBG scan if available
  * Metastatic sites: bone marrow biopsies, CT/MRI, MIBG scan
    * CR (Complete response): No tumor (primary & metastatic)
    * VGPR (Very good PR): Decreased by 90-99% (primary) & no tumor (metastatic)
    * PR (Partial response): Decreased by > 50% (primary & metastatic)
    * MR (Mixed response): > 50% reduction of any measurable lesion (primary or metastases) with < 50% reduction in any other; < 25% increase in any existing lesion
    * SD (Stable disease): No new lesions; < 50% reduction but < 25% increase in any existing lesion.
    * PD (Progressive disease): Any new lesion; increase of any measurable lesion by > 25%
Rate of tumor response (brain tumor) | 4 weeks
  - as assessed by 2-dimensional measurement (the product of the tumor's longest diameter and its longest perpendicular diameter)
  * CR: complete disappearance of all previously measurable tumors.
  * PR: greater than 50% decrease in tumor size
  * SD: less than 50% reduction in tumor size or less than 25% increase in tumor size
  * PD: greater than 25% increase in tumor size or the appearance of a new tumor
Rate of tumor response (other solid tumors) | 4 weeks
  - as assessed by The Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
  * CR: Disappearance of all target lesions.
  * PR: At least a 30% decrease in the sum of diameters of target lesions
  * SD: Neither sufﬁcient shrinkage to qualify for PR nor sufﬁcient increase to qualify for PD
  * PD: At least a 20% increase in the sum of diameters of target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea